CLINICAL TRIAL: NCT03685981
Title: Methods to Improve Preventative Care Uptake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RCT preventative care
Record Dates: First submitted 2018-08-03; First posted 2018-09-26 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incentives information provided (Experimental)
  Interventions: Other: Incentives mailer
- No incentives information provided (No Intervention)

INTERVENTIONS:
Other: Incentives mailer — Participants will receive a letter that describes the incentives provided by their health plan for following appropriate preventative care guidelines.
  Arms: Incentives information provided

SUMMARY:
The proposed study examines whether providing patients with information on the incentives for following the preventative care guidelines available through their insurance has an impact on the update of these preventative services.

ELIGIBILITY:
Inclusion Criteria:

* Patients attributed to the New York University Langone Health Clinically Integrated Network and have Medicare or Medicaid coverage (via Healthfirst) who are due for gaps in care

Exclusion Criteria:

* Any patients who do not meet the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3145 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
% of care gaps closed | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- New York University School of Medicine, New York, New York, United States